CLINICAL TRIAL: NCT06600789
Title: A Modular, Multi-Part, Multi-Arm, Phase 1/2 Study to Evaluate the Safety and Tolerability of CT7439 Alone and in Combination With Anticancer Treatments in Participants With Solid Malignancies
Brief Title: A Modular Phase 1/2 Study With CT7439 in Participants With Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Carrick Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT7439_001
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Solid Malignancies
Keywords: Solid Malignancies; Cancer Treatment; First In Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Module 1 Part A (Dose Escalation) (Experimental): Experimental: Module 1 Part A (Dose Escalation) In Part A of Module 1, a minimum of 3 participants and maximum 6 evaluable participants with locally advanced or metastatic solid tumor malignancies will receive CT7439 capsules daily in ascending dose cohorts (maximum 6 cohorts) to identify the minimally biologically active dose (MBAD), maximum tolerated dose (MTD) and/or maximum feasible dose (MFD).
  Interventions: Drug: CT7439 Capsules (0.5 mg, 1mg, 3mg)

INTERVENTIONS:
Drug: CT7439 Capsules (0.5 mg, 1mg, 3mg) — CT7439 capsules administered by mouth once a day as monotherapy with a single starting dose of 1mg in Cohort 1 on Cycle 0 Day 1, followed by a minimum 48 hours treatment -free period before continuous daily dosing in cycles of 28 days (Cycle1 onwards) until DLT or disease progression is observed.

SUMMARY:
This modular, multi-part, multi-arm, Phase 1/2, FIH study allows the evaluation of the safety and tolerability of CT7439, dosed as a monotherapy and in combination with anticancer treatment in participants with solid malignancies.

DETAILED DESCRIPTION:
This study will initially evaluate CT7439 as a monotherapy in participants with locally advanced or metastatic solid malignancies, i.e., Module 1, which includes dose escalation cohort (Part A).

- Part A of Module 1: a First-in Human dose escalation investigating the safety and tolerability of CT7439 to identify the minimum biologically active dose (MBAD) and either maximum tolerated dose (MTD) or maximum feasible dose (MFD) of CT7439 when dosed as monotherapy. SRC, consisting of study investigators and sponsor medical personnel, will be formed to monitor the safety, tolerability, PK, and PDc data during this part of the study. In Part A, cohorts (maximum 6) will be opened sequentially following review from the SRC who will make recommendations on CT7439 dosage selection for subsequent cohorts. Participants will continue to receive IMP until evidence of disease progression, unacceptable toxicities, the participant withdraws their informed consent or is withdrawn from the study, or completion of the primary study analysis.

Further cohort(s) of specific participant sub-populations may be initiated in Module 1 following approval of a protocol amendment.

ELIGIBILITY:
Core Inclusion Criteria:

* Histopathologically or cytologically confirmed diagnosis of malignant disease evaluable by RECIST v1.1
* Provision of signed written informed consent before any study-related activities, willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures and willing to permit access to stored historical tumor tissue, prior tumor radiological assessments and tumor biomarker data.
* ECOG performance status of ≤ 2 with no deterioration over the previous 2 weeks.
* Ability to take oral medications and be willing to record daily adherence to the study drug.
* Women either of non-childbearing potential, either confirmed to be post-menopausal or of childbearing potential willing to practice effective contraception for the duration of the study and for minimum 33 days after the last dose of CT7439.
* Sexually active male patients must be willing to refrain from sperm donation from the time of signing informed consent and use condoms with all sexual partners for the duration of the study and for a minimum 93 days months after the last dose of CT7439.
* Estimated life expectancy of at least 3 months, in the opinion of the investigator.

Core Exclusion Criteria:

* Prior therapy with a specific CDK12/13 inhibitor, within any timeframe prior to the first dose of CT7439.
* Participants with any other malignancy that have been active or treated within the past 3 years prior to enrolment, with the exception of cervical intraepithelial neoplasia and non-melanoma skin cancer.
* Any unresolved toxicity (except alopecia) from prior therapy of ≥ 2 Common Terminology Criteria for Adverse Events (CTCAE) Grade.
* Active or documented history of autoimmune disease.
* Any current or prior central nervous system metastases
* Active infection requiring systemic antibiotic, antifungal, or antiviral medication within 14 days prior to first dose of study drug.
* Severe or uncontrolled medical condition or psychiatric condition.
* Human immunodeficiency virus (HIV) infection, unless the study participant on anti-retroviral therapy for at least 4 weeks (28 days),and has not had an opportunistic infection within the past 12 months prior to enrollment.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, unless participant with HBV patient is on a suppressive antiviral therapy, or participant with HCV has a viral load below the limit of quantification (LoQ).
* Participant is breastfeeding or pregnant.
* Receipt of cytotoxic and/or non- cytotoxic treatment for the malignancy within 28 days before the first dose of IMP.
* Receipt of corticosteroids within 14 days before the first dose of IMP.
* Receipt of any small molecule IMP within 28 days or 5 half-lives, whichever is longer, before the first dose of IMP.
* Receipt of concomitant medication, herbal supplement, or food that is a moderate and/or strong inhibitor or inducer of CYP3A4,,strong inhibitor or inducer of CYP2D6 or P-gp or inhibitor of BCRP within 21 days before the first dose of IMP.
* Inadequate hepatic, renal and bone marrow function, receipt of a blood transfusion (blood or blood products) within 14 days before the first dose of IMP.
* Persistent (> 4 weeks) severe pancytopenia due to previous therapy rather than to disease (ANC < 0.5 × 109/L or platelets < 50 x 109/L).
* History of cardiac dysfunction and/or presence of clinically significant cardiovascular disease
* Has received a live virus vaccination within 28 days or less of planned treatment start.

Additional Module 1 inclusion criteria:

1. Clinically confirmed locally advanced or metastatic solid malignancy for which there is no potentially curative treatment option.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events will be assessed as per CTCAE v5.0. | From first dosing at Cycle 0 to until 30 days after the last dose at Cycle 6. Each cycle is 28 days
Incidence and severity of treatment emergent Laboratory Abnormalities will be assessed as per CTCAE v5.0. | From first dosing at Cycle 0 to until 30 days after the last dose at Cycle 6. Each cycle is 28 days.
Change from Baseline in Eastern Cooperative Oncology Group Cooperative Oncology Group (ECOG) Performance scale. | Screening, Cycle 0 Day 1, Cycle 1- Days 1,8,15; Cycle 2 -Days 1,15; Cycle 3 Day 1 - Cycle 6 Day 1 (each cycle 28 days); End of Treatment (within 3 days after last CT7439 dose) and End of Study (30 +/-7 days after the last CT7439 dose administration)
  ECOG has 6 levels (0 to 5). 0=Fully Active (Most Favorable Activity); 1=Restricted activity but ambulatory; 2=Ambulatory but unable to carry out work activities; 3=Limited Self-Care; 4=Completely Disabled, No self-care (Least Favorable Activity); 5=Dead.
Systolic Blood Pressure as determined by blood pressure changes from baseline in systolic blood pressure (measured in mmHg) | Screening, Cycle 0 - Days 1 and Day 2; Cycle 1 - Days 1,8,15; Cycle 2 Day 1 - Cycle 6 Day 1 (each cycle 28 days)
Diastolic Blood Pressure as determined by blood pressure changes from baseline in diastolic blood pressure (measured in mmHg) | Screening, Cycle 0 - Days 1 and Day 2; Cycle 1 - Days 1,8,15; Cycle 2 Day 1 - Cycle 6 Day 1 (each cycle 28 days)
Heart Rate as determined by heart rate changes from baseline in beats per minute | Screening, Cycle 0 - Days 1 and Day 2; Cycle 1 - Days 1,8,15; Cycle 2 Day 1 - Cycle 6 Day 1 (each cycle 28 days)
Body Temperature. as determined by body temperature changes from baseline in Celsius or Fahrenheit | Screening, Cycle 0 - Days 1 and Day 2; Cycle 1 - Days 1,8,15; Cycle 2 Day 1 - Cycle 6 Day 1 (each cycle 28 days)
Respiratory Rate as determined by respiratory rate changes from baseline in breaths per minute | Screening, Cycle 0 - Days 1 and Day 2; Cycle 1 - Days 1,8,15; Cycle 2 Day 1 - Cycle 6 Day 1 (each cycle 28 days)
Oxygen Saturation as determined by changes from baseline in % | Screening, Cycle 0 - Days 1 and Day 2; Cycle 1 - Days 1,8,15; Cycle 2 Day 1 - Cycle 6 Day 1 (each cycle 28 days)
Change from Baseline in 12-lead Electrocardiogram (ECG): Heart Rate | From baseline to end of Cycle 6. Each cycle is 28 days
Change from Baseline in 12-lead Electrocardiogram (ECG): PR interval | From baseline to end of Cycle 6. Each cycle is 28 days
Change from Baseline in 12-lead Electrocardiogram (ECG): QRS complex | From baseline to end of Cycle 6. Each cycle is 28 days
Change from Baseline in 12-lead Electrocardiogram (ECG): QT intervals | From baseline to end of Cycle 6. Each cycle is 28 days
Change from Baseline in 12-lead Electrocardiogram (ECG): QTcF intervals (QT Interval Corrected by the Fridericia Formula) | From baseline to end of Cycle 6. Each cycle is 28 days
Module 1 Part A additional primary outcome measures: Maximum tolerated dose (MTD) determination | Up to 28 days after the first dose of CT7439
  Maximum tolerated dose (MTD) defined as the highest dose level at which ≤ 1/6 participants experience DLT in the first cycle. A minimum of 6 participants must be enrolled at the MTD level

SECONDARY OUTCOMES:
CT7439 PK Plasma exposure: Cmax | PK urine exposure Cmax: At the end of Cycle 0 Day 1 (cycle 0 is 2 days)
  Maximum PK Plasma concentrations and PK parameters for CT7439
CT7439 PK plasma exposure: C-trough | Cycle 0 Day 2, Cycle 1 - Days 1, 8, 15; Cycle 2 Day 2; on Cycle 3 day 1 and upwards on Day 1 of every other cycle (each cycle is 28 days)
  CT7439 PK plasma parameters pre-dose
Changes in CT or MRI tumor imaging to monitor anti-tumor activity | Screening, Cycles 3 Day 1 to Cycle 6 Day 1 (28 days each cycle) and End of Module/ End of Treatment visit (within 3 days after last CT7439 dose)
  the imaging method of CT or MRI will be used at each subsequent visit
CT7439 PK urine exposure: Cmax | At Cycle 0, Day 1. Cycle 0 Day 1 is 24 hours.
  CT7439 PK concentration in urine
Module 1 Part A additional secondary outcome measures - determination of recommended Phase 2 Dose (RP2D) and minimally biologically active dose (MBAD) of CT7439 when administered as monotherapy | from cohort 1 to cohort 6. (each cohort is 6 cycles , each cycle is 28 days)
  the CT7439 MBAD is defined as the dose level that will show / achieve a proof of mechanism (PoM) ;a partial or complete RECIST v1.1 assessed response in at least one participant; a clinically significant reduction (in the opinion of the safety review committee (SRC), compared to baseline, in a tumor-specific marker measured in at least one participant
Module 1 Part A additional secondary outcome measures - Incidence of Dose Limited Toxicities (DLT) | At end of Cycle 1 (each cycle is 28 days)
  number of safety events that are not clearly due to the underlying disease or extraneous causes lead to death, or discontinuation of drug treatment due to non-hematological toxicities (Grade 3 or higher) or hematological toxicities (Grade 3 or higher)
Module 1A secondary outcome measures- Renal clearance | Screening, Cycle 0 Day 1, Cycle 1 - Day 1,8,15, Cycle 2 - Day 1,15; Cycle 3 - Cycle 6 (28 day each cycle), End of Module/ End of Treatment (within 3 days after last CT7439 dose)
  Serum Chemistry creatinine clearance
Module 1A secondary outcome measures - Pharmacodynamic evidence of the downstream effects of target engagement | Screening; Cycle 0 Day 1; Cycle 1 - Day 1, 8 and 15; Cycle 2- Cycle 6 (28 day each cycle) - Day 1; and EOT visit
  Whole blood RNA assay
Module 1A secondary outcome measures - Incidence and prevalence of adverse events (AE) resulting in treatment withdrawal | From 1st dose of IMP administration at Cycle 0 Day 1 throughout treatment Cycles 1, Cycle 2 - Cycles 6 ( each cycle 28 days) and until End of Treatment (within 3 days of last CT7439 dose) and End of Study (30+/- 7 days after the last CT7439 dose)
  number of adverse events leading to investigational medicinal drug (IMP) withdrawal
Module 1A secondary outcome measures - Best overall response (BOR) | Up to 24 weeks
  BOR defined as the best response recorded from the randomization start until disease progression or death due to any cause
Module 1A Overall response rate (ORR) | Up to 24 weeks
  ORR defined as the proportion of participants who achieved a complete response (CR) or partial response (PR) as per RECIST Version 1.1
Module 1A Duration of Response (DOR) | Up to 24 weeks
  DOR defined as the time from the date of first documentation of objective tumor response (CR or PR) to the first documented objective tumor progression per RECIST version 1.1 or censored as defined for PFS
Module 1A PFS (Progression-free survival) assessment | Up to 18 months
  PFS defined as the time from the first dose of IMP to the date of the first documentation of objective progression of disease (PD) per RECIST version 1.1

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Research site 03, Dallas, Texas
  - Research site 01, San Antonio, Texas
  - Research site 02, Fairfax, Virginia
- United Kingdom (3):
  - Research site 05, Manchester
  - Research site 04, Oxford
  - Research site 06, Sutton

IPD SHARING:
Plan to Share IPD: No